CLINICAL TRIAL: NCT05087121
Title: A Pilot Study of Cognitive Behavioral Therapy - Insomnia (CBT-I) Among Professional Firefighters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pacific University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1684868-2
Record Dates: First submitted 2021-06-28; First posted 2021-10-21 (Actual); Last update posted 2022-12-01 (Actual); Status verified 2022-09

CONDITIONS: Insomnia; Shift-Work Related Sleep Disturbance
Keywords: Sleep; Firefighter; CBT-I
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Two-group design in which eligible participants are randomized via permuted block, with a block size of seven, to either the intervention (CBT-I-F) condition or a no intervention control condition. Unequal allocation to groups based on 60:40 split, intervention:control. Randomization stratified according to gender identity.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Cognitive Behavioral Therapy for Insomnia for Firefighters (CBT-I-F) [Treatment Group] (Experimental): The Cognitive Behavioral Therapy for Insomnia for Firefighters (CBT-I-F) is a 6-week training course that focuses on mitigating poor sleep quality and promoting the adoption of behaviors conducive to quality sleep. This course includes modules on developing habits conducive to better sleep, adapting variable bedroom environments, and establishing techniques to reduce worry and frustration around falling asleep while recognizing and working through barriers unique to the career of firefighting.
  Interventions: Behavioral: Cognitive Behavioral Therapy for Insomnia for Firefighters (CBT-I-F); Device: Fitbit Inspire HR Wrist Worn Device (NCT04176926)
- No Intervention Control Group (No Intervention): Non-Intervention Control Group (NIC) will not receive training during the course of the study, but will be offered the opportunity to receive training after the study ends.

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy for Insomnia for Firefighters (CBT-I-F) — The Cognitive Behavioral Therapy for Insomnia for Firefighters (CBT-I-F) 6-week training course has been derived from existing Cognitive Behavioral Therapy for Insomnia (CBT-I) group therapy protocols. Participants in this intervention will receive psychoeducation on sleep and practice skills standard of CBT-I including, stimulus control techniques, sleep restriction, counter-arousal skills, cognitive restructuring, sleep hygiene, goal setting, and relapse prevention skills. Weekly sessions will include discussions regarding difficulties specific to occupational barriers and how to mitigate the impact of occupational requirements on sleep quality.
  Other Names: CBT-I; Cognitive Behavioral Therapy - Insomnia
  Arms: Cognitive Behavioral Therapy for Insomnia for Firefighters (CBT-I-F) [Treatment Group]
Device: Fitbit Inspire HR Wrist Worn Device (NCT04176926) — The Fitbit Inspire HR wrist worn device will be worn by eligible participants throughout the duration of the intervention and for two weeks following completion of the 6-week intervention to collect objective data on enduring sleep changes. This device is an FDA-registered medical device that is not the object of investigation and is being used "on label" only to gather data.
  501(K) Number: K200948 Device Name: Fitbit ECG App Regulation Number: 870.2345 Classification Product Code: QDA Clinical Trials: NCT04176926
  Arms: Cognitive Behavioral Therapy for Insomnia for Firefighters (CBT-I-F) [Treatment Group]

SUMMARY:
The primary aim of this study is to investigate the feasibility, acceptability, and preliminary efficacy of an adapted Cognitive Behavioral Therapy - Insomnia (CBT-I) intervention in improving sleep in a firefighter population.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, participants will be randomized to the intervention group (group to receive CBT-I) or the no-intervention control group. All participants in the study will complete three assessment visits; one prior to the start of the intervention, one immediately following the 6-week intervention, and one 3-months post-intervention. The intervention group will engage in 6-weeks of CBT-I training aimed at targeting sleep and sleep-related concerns faced as a result of occupational considerations.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* full-time professional firefighter
* At least 18 years of age
* A global Pittsburgh Sleep Quality Index score ≥ 5 (Grandner et al., 2006)
* Be willing and able to participate in all study activities including pre-, post-, and 3-month follow up assessments and 6-weeks of the CBT-I intervention
* Agree to random assignment to one of two conditions (treatment or control group)
* Have access to an email account
* Be willing to wear the Fitbit Inspire HR device throughout the duration of the intervention and for two weeks following completion of the 6-week intervention

Exclusion Criteria:

* Endorsement of prior involvement in formal CBT-I interventions
* Unwillingness to give written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2021-02-16 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Change in Scores on the Pittsburgh Sleep Quality Index (PSQI) | Baseline (i.e., pre-intervention), 6 weeks (i.e., post-intervention), 18 weeks (i.e., 3-month follow-up)
  The Pittsburgh Sleep Quality Index (PSQI) is a self-report questionnaire designed to assess sleep quality and sleep disfunction throughout the previous month. Global scores range between 0-21 with higher scores indicating greater sleep dysfunction.
Total Sleep Time Change as Measured by Actigraphy in the Fitbit Inspire HR | Baseline (i.e., pre-intervention), 6 weeks (i.e., post-intervention)
  Fitbit Inspire HR wrist worn devices will be used to assess mean sleep patterns and sleep-related activity. The Fitbit Inspire HR may be worn consistently for up to 5-days and records wrist movement and heart rate variability to estimate sleep onset, waking, and sleep stages without need for the wearer to actively manipulate the device.
Feasibility as measured by attendance, attrition, and adherence to intervention components. | From intervention Week 1 to intervention Week 6
  Feasibility will be measured via attendance, attrition rates, and completion of sleep diaries Participant weekly CBT-I attendance will be tracked and analyzed based upon average percentage of total number of sessions attended. Adherence to intervention components will be tracked via compliance with recommendations for the previous week. After each session, sleep diaries for that week will be examined by research assistants and recorded dichotomously as to whether "Yes, the participant was adherent" or "No, the participant was not adherent". An adherence percentage will be calculated.
Acceptability as measured by mean acceptability ratings on four Likert-style questions. | 6 weeks (i.e., post-intervention)
  Acceptability will be assessed using four self-report questions derived from similar studies, and calculated via mean acceptability ratings on a scale of 0-6. These items will include the degree to which the participant liked the program, whether they found the home practice/requirements reasonable, whether they would recommend the program, and whether they would take the program again in the future. Each item is responded to on a 7-point Likert-type scale ranging from 0 to 6, with higher scores indicating greater acceptability.

SECONDARY OUTCOMES:
Depression, Anxiety, and Stress as Measured Through the Depression, Anxiety, and Stress Scales 21 (DASS-21). | Baseline (i.e., pre-intervention), 6 weeks (i.e., post-intervention), 18 weeks (i.e., 3-month follow-up)
  The Depression, Anxiety, Stress Scales 21-item measure (DASS-21) measures self-report ratings of depression, anxiety, stress symptoms. Items are responded to on a 4-point Likert-type scale ranging from 0 (Did not apply to me at all) and 3 (Applied to me very much or most of the time). Scores range between 0 and 120 for the DASS-21 total score. Higher scores indicate a greater severity of depression, anxiety, and stress.
PTSD as Measured Through the PTSD Checklist for DSM-5 (PCL-5) | Baseline (i.e., pre-intervention), 6 weeks (i.e., post-intervention), 18 weeks (i.e., 3-month follow-up)
  The PTSD Checklist for DSM-5 (PCL-5) measures self-reported PTSD symptoms. Items are responded to on a 5-point Likert-type scale ranging between 0 (Not at all) to 4 (Extremely) with higher scores indicating greater severity of PTSD symptoms. Items are summed to create a total score ranging between 0-80 and scores greater than 33 indicate probable PTSD.
General Health as Measured Through the Medical Outcomes Study 12-item Short-Form Survey (SF12v2) | Baseline (i.e., pre-intervention), 6 weeks (i.e., post-intervention), 18 weeks (i.e., 3-month follow-up)
  The Medical Outcomes Study 12-item Short-Form Survey (SF12v2) measures self-reported general health. The SF12v2 is a 12-item self-report that contains eight subscales: physical functioning, role-physical (i.e., role limitations related to physical health), bodily pain, general health, vitality, social functioning, role-emotional (i.e., emotional problems resulting in role limitations), and mental health. Higher scores indicate more favorable states of health.
Family Functioning as Measured Through the McMaster Family Assessment Device - General Functioning Scale (FAD-GFS) | Baseline (i.e., pre-intervention), 6 weeks (i.e., post-intervention), 18 weeks (i.e., 3-month follow-up)
  The McMaster Family Assessment Device - General Functioning Scale (FAD-GFS) measures self-reported family functioning. The FAD-GFS is a 12-item self-report subscale of the larger 60-item FAD measure, that assesses overall health and pathology of the family. Items on the FAD-GFS are responded to on a 4-point Likert-type scale ranging between 1 (Strongly Agree) and 4 (Strongly Disagree). Higher total scores indicate more problematic family functioning.
Vigilant Attention as Measured Through the Psychomotor Vigilance Task (PVT). | Baseline (i.e., pre-intervention), 6 weeks (i.e., post-intervention), 18 weeks (i.e., 3-month follow-up)
  The Psychomotor Vigilance Task (PVT) is a continuous performance task commonly used to objectively assess sleep-related cognitive deficits in vigilant attention. The PVT, administered remotely via Inquisit Web software (Millisecond Software LLC, US) will be used in this study. Inter-stimulus intervals are set to vary randomly between 2-10 seconds and subjects are to respond as quickly as possibly by clicking the mouse to stimuli flashed on the screen. Higher scores indicate slower response times and greater number of errors.
Fidelity of Intervention Protocol Across Sessions | 6 weeks (i.e., post-intervention)
  Fidelity will be assessed to ensure therapist adherence to the intervention protocol in each session. An adherence measure of covered session topics, covered activities, and global instructor skill in presenting material will be used to for each weekly session. Sessions will be audio recorded and two research assistants will independently rate each item regarding covered session topics and covered activities on a 3-point Likert-style scale ranging from 0-2 (0 = not present, 1 = somewhat present, 2 = fully present), and global instructor skill in presenting the material will also be rated on a 3-point Likert-style scale ranging from 0-2 (0 = none, 1 = minimal, 2 = adequate). Higher scores indicate better fidelity.

CONTACTS AND LOCATIONS:
Overall Officials: Kaylie A Green, M.S., Principal Investigator — Pacific University; Michael Christopher, Ph.D., Study Chair — Pacific University
Locations (1):
- Pacific University, Forest Grove, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
We are committed to advancing knowledge in the scientific community and the role that data sharing takes in this endeavor. We agree to share all final, de-identified research data as broadly as possible to the extent consistent with applicable laws, regulations, rules, and policies. As requested, aggregate data in the form of summary statistics and tables will be shared, with description of analytical methods used. Data requests will be carefully evaluated to insure that the data are sought for scientifically-sound reasons, that the individual requesting the data is professionally qualified, and that the data to be shared are properly de-identified so as to protect the rights of participants. When de-identifying the data, care will be taken to remove identifiers while maintaining the scientific integrity of the data. Removing both direct and indirect identities will be undertaken to insure that even deductive disclosure of identity is unlikely.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: The data generated in this study will be presented at regional, national, and international conferences and published in peer-reviewed journals in a timely fashion. All final peer-reviewed manuscripts that arise from this proposal will be submitted to the digital archive PubMed Central.
Access Criteria: Data sharing agreements will be required to ensure that the data will be used only for research purposes and will not be transferred to others without first notifying and receiving permission. The data will be stored in SPSS format by the multiple principal investigators and, following completion of a data sharing agreement, will be distributed directly by one of the multiple principal investigators via electronic file.

DOCUMENTS (1):
  • Informed Consent Form (2021-02-16): https://cdn.clinicaltrials.gov/large-docs/21/NCT05087121/ICF_000.pdf